CLINICAL TRIAL: NCT06042985
Title: Comparison of the Absorption of Calcium Citrate and Calcium Carbonate in Patients With an RYGB, LSG, and OAGB A Double-blind, Randomized Cross-over Trial
Brief Title: Comparison of the Absorption of Calcium Citrate and Calcium Carbonate in Patients With an RYGB, LSG, and OAGB
Acronym: CALCOR-RSO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Principal Investigator, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AU-calcium-rct-23
Record Dates: First submitted 2023-08-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Calcium Citrate Absorption; Calcium Carbonate Absorption
Keywords: Calcium Citrate; bariatric surgery; Absorption; Calcium Carbonate
MeSH Terms: interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: In a double-blind-randomization procedure, surgeons, the research team, the laboratory, and the statistical analysis team will be blinded; the patient has no influence and not necessary to be blind.
Who Masked: Participant
Masking Description: All the patients will be used in a cross-over study design. The same patient will be using study drugs A or B and switching in the study to the other drug.
  7 days period will be applied for any wash-out or possible carry-over effect.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RYGB arm: calcium citrate and calcium carbonate (Active Comparator): The absorption effect between calcium citrate and calcium carbonate in patients with a RYGB
  Interventions: Drug: The absorption effect between calcium citrate and calcium carbonate
- LSG arm: calcium citrate and calcium carbonate (Active Comparator): The absorption effect between calcium citrate and calcium carbonate in patients with a LSG
  Interventions: Drug: The absorption effect between calcium citrate and calcium carbonate
- OAGB arm: calcium citrate and calcium carbonate (Active Comparator): The absorption effect between calcium citrate and calcium carbonate in patients with a OAGB
  Interventions: Drug: The absorption effect between calcium citrate and calcium carbonate

INTERVENTIONS:
Drug: The absorption effect between calcium citrate and calcium carbonate — Elemental Calcium citrate supplementation will significantly improve patients' absorption after BMS in all cases.
  Other Names: Elemental Calcium citrate; Elemental Calcium Carbonate; Chewable tablets

SUMMARY:
The precise impact of calcium absorption in relation to RYGB, SG, and OAGB remains under-researched in terms of statistical power and the diversity of BMS procedures considered. Therefore, this presents a critical area for future investigation to improve patient outcomes in BMS.

DETAILED DESCRIPTION:
Calcium, predominantly absorbed in the duodenum and proximal jejunum, relies heavily on vitamin D and an acidic environment to facilitate absorption. With the increasing prevalence of bariatric metabolic surgery (BMS) procedures and their malabsorptive effects, the likelihood of fat-soluble vitamin malabsorption becomes heightened. This stems from bypassing the stomach, key absorption sites in the intestine, and the inefficient mixing of bile salts.

BMS is often associated with several bone metabolism disorders, including the acceleration of bone remodeling and turnover, bone loss, and decreased bone mineral density (BMD). Postoperative calcium supplementation can mitigate this bone loss over time. For instance, a study demonstrated the beneficial effect of calcium citrate following Roux-en-Y gastric bypass (RYGB). However, the study's statistical power was insufficient; thus, the BMS field still awaits further conclusive and robust research to establish definitive guidelines, which was highlighted in another study.

Moreover, substantial changes in gut hormones, such as peptide YY (PYY), glucagon-like peptide-1, and ghrelin, have been observed following RYGB, sleeve gastrectomy (SG), and One Anastomosis Gastric Bypass (OAGB). While these hormonal changes are typically associated with BMS's numerous positive metabolic benefits, they may also contribute to bone loss.

Consequently, the precise impact of calcium absorption in relation to RYGB, SG, and OAGB remains under-researched in terms of statistical power and the diversity of BMS procedures considered. Therefore, this presents a critical area for future investigation to improve patient outcomes in BMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years old
* After BMS surgery who had an RYGB, SG, or OAGB operation at least 12 months before the study.
* Patients will be selected at random from the hospital's electronic patient system.

Exclusion Criteria:

* Patients on antacids during the study
* Patients onH2 receptor antagonists during the study
* Patients on proton pump inhibitors during the study
* Patients with a previous oophorectomy,
* Liver disease,
* Renal disease,
* Hypercalcemia,
* Hyperthyroidism,
* Hypothyroidism who require levothyroxine supplementation (Levothyroxine forms complexes with calcium)
* Parathyroid disorders
* Use of diuretics,
* Use of calcitonin,
* Use of corticosteroids,
* Use of anabolic steroids,
* Use of anticonvulsants within three months of the study
* Heavy smokers (>10 cigarettes/day)
* Abusing alcohol (>70 ml/day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Elemental Calcium effects in blood serum (Peak Plasma Concentration (Cmax)) | 8 hours
  In patients who have undergone bariatric surgery and are receiving elemental calcium supplementation in the form of citrate or carbonate, we observe variations in their blood serum with peak concentrations (Cmax)
  These changes provide insights into how effectively the body absorbs and utilizes calcium following supplementation.
Elemental Calcium effects in Urine excretion (time curve (AUC)) | 8 hours
  In patients who have undergone bariatric surgery and are receiving elemental calcium supplementation in the form of citrate or carbonate, we observe variations in their cumulative excretion of urinary calcium over time (AUC).
  These changes provide insights into how effectively the body absorbs and utilizes calcium following supplementation.
Elemental Calcium effects in blood serum (Area under the plasma concentration) | 8 hours
  In patients who have undergone bariatric surgery and are receiving elemental calcium supplementation in the form of citrate or carbonate, we observe variations in their blood serum with Area under the plasma concentration (AUC)
  These changes provide insights into how effectively the body absorbs and utilizes calcium following supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: M Hany Ashour, MD, Principal Investigator — Alexandria University
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after study completed, for 15 years
Access Criteria: contact study PI

REFERENCES:
- [Background] Allied Health Sciences Section Ad Hoc Nutrition Committee; Aills L, Blankenship J, Buffington C, Furtado M, Parrott J. ASMBS Allied Health Nutritional Guidelines for the Surgical Weight Loss Patient. Surg Obes Relat Dis. 2008 Sep-Oct;4(5 Suppl):S73-108. doi: 10.1016/j.soard.2008.03.002. Epub 2008 May 19. No abstract available. PMID 18490202
- [Background] Mechanick JI, Apovian C, Brethauer S, Garvey WT, Joffe AM, Kim J, Kushner RF, Lindquist R, Pessah-Pollack R, Seger J, Urman RD, Adams S, Cleek JB, Correa R, Figaro MK, Flanders K, Grams J, Hurley DL, Kothari S, Seger MV, Still CD. CLINICAL PRACTICE GUIDELINES FOR THE PERIOPERATIVE NUTRITION, METABOLIC, AND NONSURGICAL SUPPORT OF PATIENTS UNDERGOING BARIATRIC PROCEDURES - 2019 UPDATE: COSPONSORED BY AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS/AMERICAN COLLEGE OF ENDOCRINOLOGY, THE OBESITY SOCIETY, AMERICAN SOCIETY FOR METABOLIC & BARIATRIC SURGERY, OBESITY MEDICINE ASSOCIATION, AND AMERICAN SOCIETY OF ANESTHESIOLOGISTS - EXECUTIVE SUMMARY. Endocr Pract. 2019 Dec;25(12):1346-1359. doi: 10.4158/GL-2019-0406. Epub 2019 Nov 4. PMID 31682518
- [Background] Tondapu P, Provost D, Adams-Huet B, Sims T, Chang C, Sakhaee K. Comparison of the absorption of calcium carbonate and calcium citrate after Roux-en-Y gastric bypass. Obes Surg. 2009 Sep;19(9):1256-61. doi: 10.1007/s11695-009-9850-6. Epub 2009 May 13. PMID 19437082
- [Background] Smelt HJ, Pouwels S, Smulders JF. The Clinical Dilemma of Calcium Supplementation After Bariatric Surgery: Calcium Citrate or Calcium Carbonate That Is the Question? Obes Surg. 2016 Nov;26(11):2781-2782. doi: 10.1007/s11695-016-2346-2. No abstract available. PMID 27558620
- [Result] Schafer AL, Weaver CM, Black DM, Wheeler AL, Chang H, Szefc GV, Stewart L, Rogers SJ, Carter JT, Posselt AM, Shoback DM, Sellmeyer DE. Intestinal Calcium Absorption Decreases Dramatically After Gastric Bypass Surgery Despite Optimization of Vitamin D Status. J Bone Miner Res. 2015 Aug;30(8):1377-85. doi: 10.1002/jbmr.2467. Epub 2015 May 21. PMID 25640580